CLINICAL TRIAL: NCT03385798
Title: Endo-GIA Versus Endowrist Stapler in Intracorporeal Urinary Diversion in Robotic Assisted Radical Cystectomy
Acronym: EGIAES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jørgen Bjerggaard Jensen (Other)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, MD, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFE-1-10-72-78-17
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Bladder Cancer
Keywords: Endo-GIA Stapler; Endowrist Stapler
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endo-GIA (Active Comparator)
  Interventions: Procedure: Endo-GIA
- Endo-wrist (Experimental)
  Interventions: Procedure: Endowrist

INTERVENTIONS:
Procedure: Endowrist — Anastomosis made by Endowrist
  Arms: Endo-wrist
Procedure: Endo-GIA — Anastomosis made by Endo-GIA
  Arms: Endo-GIA

SUMMARY:
The study is a randomized clinical trial (RCT) including patients undergoing robotic assisted cystectomy with intracorporeal ileal conduit at four large university hospitals in Denmark.

If included, the patients will be randomized 1:1 to two study arms: 1) Standard arm with current procedure where intracorporeal bowel anastomosis is performed with the 60 mm EndoGIA stapler, or 2) Experimental arm where the bowel anastomosis will be performed totally robotic with the Endowrist Intuitive robotic stapler with 2 subsequent elongated 45 mm magazines for the side-to-side anastomosis.

Primary outcome will be postoperative bowel function where a better bowel recovery is anticipated in the experimental Endowrist arm whereas serious complications are expected to be non-inferior to the current standard.

DETAILED DESCRIPTION:
Cystectomy with urinary diversion is the standard treatment of muscle invasive and high risk non-muscle invasive bladder cancer. During cystectomy, a urinary diversion is constructed from a bowel segment. Restoration of the intestinal continuity is therefore an obligate part of the procedure.

In Denmark, approximately 400 radical cystectomies are performed yearly with the majority of procedures performed as a laparoscopic robot assisted procedure. This includes urinary diversion by means of intracorporeal procedure.

During current standard intracorporeal urinary diversion, an Endo-GIA stapler is handled by the assisting surgeon and not by the main surgeon as the Endo-GIA stapler is not integrated into the robot.

The traditional Endo-GIA anastomosis is made as a side-by-side anastomosis with two 60 mm magazines: one for the side-to-side anastomosis and one for closing the end.

Any reduction in the lumen of the anastomosis will clinically affect post-operative bowel function. It is known that at all cystectomy patients have intestinal paralysis / lack of normal bowel function in the first days postoperatively. It is thus plausible that a wider anastomosis will be able to reduce the duration of this in favor of the patient's post-operative nutrition, postoperative length of stay and convalescence.

A stapler integrated in the robot (Endowrist stapler from Intuitive) is available. This has several advantages: it is operated by the robotic surgeon and not by the assistant, it is more flexible, and faster mobility. These advantages provide the possibility of precisely removing a minimal intestinal segment by the final transverse stapling. The biggest disadvantage of the robot-operated Endowrist staple is that it is not available in a 60 mm version but only in 45 mm, thus giving only an anastomosis of approximately the same lumen as using a 60 mm Endo-GIA staple but not better.

An opportunity to make a more spacious anastomosis would be to "prolong" the longitudinal stapling as to the side-to-side anastomosis between the intestinal segments. This requires precise and coordinated handling of bowel graspers and staplers to make a complete elimination of the risk of anastomosis leakage, which in this respect is an advantage of robot-operated staples with the Endowrist stapler rather than an assistant handled stapler with Endo-GIA.

Both Endo-GIA and Endowrist stapler are approved for clinical use according to the procedures described.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* The ability to understand Danish orally and in writing
* undergoing robotic assisted cystectomy with intracorporeal ileal conduit

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative bowel function | 90 days
  Primary outcome will be postoperative bowel function where a better bowel recovery is anticipated in the experimental Endowrist arm whereas serious complications are expected to be non-inferior to the current standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choy PY, Bissett IP, Docherty JG, Parry BR, Merrie A, Fitzgerald A. Stapled versus handsewn methods for ileocolic anastomoses. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD004320. doi: 10.1002/14651858.CD004320.pub3. PMID 21901690
- [Background] Korolija D. The current evidence on stapled versus hand-sewn anastomoses in the digestive tract. Minim Invasive Ther Allied Technol. 2008;17(3):151-4. doi: 10.1080/13645700802103423. PMID 18609000
- [Background] Chen C. The art of bowel anastomosis. Scand J Surg. 2012;101(4):238-40. doi: 10.1177/145749691210100403. PMID 23238497
- [Background] Dal Moro F, Haber GP, Wiklund P, Canda AE, Balbay MD, Stenzl A, Zattoni F, Palou J, Gill I, Catto JW. Robotic intracorporeal urinary diversion: practical review of current surgical techniques. Minerva Urol Nefrol. 2017 Feb;69(1):14-25. doi: 10.23736/S0393-2249.16.02780-6. Epub 2016 Aug 31. PMID 28009143
- [Background] Russell KW, O'Holleran BP, Bowen ME, Mone MC, Scaife CL. The Barcelona Technique for Ileostomy Reversal. J Gastrointest Surg. 2015 Dec;19(12):2269-72. doi: 10.1007/s11605-015-2929-6. Epub 2015 Sep 4. PMID 26341822
- [Background] Jensen JB, Pedersen KV, Olsen KO, Bisgaard UF, Jensen KM. Mini-laparotomy approach to radical cystectomy. BJU Int. 2011 Oct;108(7):1125-30. doi: 10.1111/j.1464-410X.2010.09958.x. Epub 2011 Jan 11. PMID 21223476
- [Background] Ducrotte P, Causse C. The Bowel Function Index: a new validated scale for assessing opioid-induced constipation. Curr Med Res Opin. 2012 Mar;28(3):457-66. doi: 10.1185/03007995.2012.657301. Epub 2012 Feb 16. PMID 22236136